CLINICAL TRIAL: NCT05986175
Title: The Effect of Motor Imagery Training in Addition to Core Stabilization Exercises on Core Performance, Balance, Functional Capacity, and Quality of Life in Healthy Adolescents Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: buhucgun02
Record Dates: First submitted 2023-07-04; First posted 2023-08-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Adolescent
Keywords: Motor Imagery Training; Core Stabilization Exercises; Adolescent

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery Training Group (Experimental): The Motor Imagery Training Group will receive motor imagery training in addition to Jeffreys' core (body) stabilization training protocol.
  Interventions: Other: Motor Imagery Training; Other: Core Stabilization Exercises
- Core Stabilization Exercises Group (Active Comparator): The Core Stabilization Exercises Group will receive only Jeffreys' core (body) stabilization training protocol.
  Interventions: Other: Core Stabilization Exercises

INTERVENTIONS:
Other: Motor Imagery Training — The motor imagery training will be given with an audio recording containing 15 minutes of motor imagery training. The protocol will be administered by a physiotherapist 3 times a week for 8 weeks.
  Arms: Motor Imagery Training Group
Other: Core Stabilization Exercises — Jeffreys' Core (body) Stabilization Exercises will be implemented. The protocol consists of exercises that progress gradually from the first level to the third level. The first level consists of static contraction training on a stable surface; the second level is dynamic training on stable surfaces; and the third level is dynamic and resistant training on an unstable surface. Each session is scheduled to last 45 minutes, with 5 minutes of heating and 5 minutes of cooling exercises. The protocol will be administered by a physiotherapist 3 times a week for 8 weeks.

SUMMARY:
Adolescence is the period in which a person grows and develops the fastest, covering the transition from childhood to maturity. Compared to sedentary adolescents who regularly exercise, there were significant differences in levels of functional capacity, cognitive function, and quality of life. The balance that shows significant development in the adult period, if not sufficiently developed, results in a lack of proper balance during movements, making individuals exposed to injuries.

A strong "core" area is needed to ensure the stabilization of the whole body and increase functional capacity. In the studies carried out, the "core" exercise programs resulted in increased lumbopelvic stability, improved small and large muscle strength, and increased body control and balance.

Motor imagery is defined as the resurrection of movement in the mind before movement occurs. For individuals with health or health-related problems, it has been found that the implementation of imaging tasks is beneficial, either alone or in addition to physical practice and that similar brain regions are activated during the performance of the movement and imaging the movement.

56 healthy girls will be included in our study. The participants will be randomly divided into 2 groups, including 28 control groups and 28 training groups. The core performance will be assessed with the Modified Push-Up Test and Sit-Up Test. The Flamingo test will be used to assess static balance and the Y test will be used to assess dynamic balance. Quality of life will be assessed with the Pediatric Quality of Life Questionnaire (PedsQL) for adolescents aged 13-18 years. Functional capacity will be assessed with the 6-Minute Walk Test. Exercise Readiness Questionnaire will be used to measure exercise readiness. The Movement Imagery Questionnaire-Revised (MIQ-R) form will be used for motor imagery; the Vividness of Motor Imagery Questionnaire (VMIQ) will be used for clarity and vividness of motor imagery. During the motor imagery training, heart rate will be measured to determine whether the participant performs the imagery correctly. In addition to all of these assessments, the values of Heart Rate, Blood Pressure, Saturation, Dyspnea, and Fatigue Levels (Modified Borg Dyspnea and fatigue scales) will be recorded. The control group will be subject to Jeffreys' core (body) stabilization training protocol. The training group will receive engine simulation training in addition to Jeffreys' core (body) stabilization training protocol. The control group and the training group will implement training programs with a physiotherapist 3 times a week for 8 weeks. All assessments will be repeated before and after the 8-week training program.

The aim of the present study is to investigate the effect of motor imagery training given in addition to core stabilization training on core performance, balance, functional capacity, and quality of life in healthy adolescent girls.

ELIGIBILITY:
Inclusion Criteria:

* Being between 10 and 19 years old
* Having no barriers to exercise according to Activity Readiness Questionare for Everyone (PAR-Q+)
* To get a valid score from Vividness of Imagery Questionnaire (VMIQ)
* To volunteer to participate in the study

Exclusion Criteria:

* Having had any neurological and orthopedic injury in the last 1 year
* Having a history of any vestibular-visual disease that may affect balance
* Having a history of any disease that may cause disability or systemic problems during exercise

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Core Performance | 5 -10 minutes
  The Modified Push-Up Test will be used to assess the measure the strength and endurance of the upper extremity. The participant is positioned face-to-face on the arm, the knees and elbows are folded, and the hands are in the shoulder line and next to the body. The individual is asked to lift his upper body and body from the ground, bringing his elbow to extension without disturbing the flexion in his knees.
Core Performance | 5 -10 minutes
  The Sit-Up Test will be used to assess the core performance. The knees are bent, the feet are on the ground, and the arms lie on the back in a crossed position on the chest. The participant is asked to raise his back to 90 degrees from the ground within 30 seconds and then take the starting position again. Supporting the feet helps to move. The movement starts when you are on the back, and when you get to the same position, 1 is counted again.
Balance | 10 - 15 minutes
  The Flamingo Test will be used to assess the duration of static balance on a single foot. The participant is held on a wooden platform with a length of 50 cm, holding one foot back on the platform with the hand on the same side, and holding it like a flamingo. Run to balance with the remaining free arm, the test practitioner holds his arm to balance and starts the period when he leaves his arm. The disturbance of the position is stopped when the foot moves and the hand leaves the leg, and the time is continued again when the participant is ready. The period until the loss of balance is calculated, and the number of losses, disruptions, or falls within 60 seconds is recorded during balancing. Participants who drop more than 15 in the first 30 seconds are awarded zero points.
Balance | 5 - 10 minutes
  Y-balance test which is a modification of the Star Excursion Balance Test (SEBT) will be used to assess the balance. The participant, standing on his preferred foot on a 50 cm long wooden platform on a 4 cm high and 3 cm wide balance platform (flamingo balance test), tries to stay in balance for 1 minute by bending the other foot from the knee, pulling it to the hip, and holding it with the same hand on the same side.
Functional Capacity | 15-20 minutes
  The 6-minute walking test will be used to assess the functional capacity. Participants will be recorded in a 30-meter straight corridor for 6 minutes at their own walking speed, as fast as possible but without running. The walking distance will be recorded in meters.
Movement Imagery Ability | 25 - 30 minutes
  The Motion Imaging Survey - Revised Second Edition will be used to assess the visual and kinesthetic imaging skills. It consists of a total of 14 elements, including visual and kinesthetic imaging. Scores that can be obtained from the scale range between 14-98. High scores mean that the level of visual imagery is also high.
Movement Imagery Ability | 15 - 20 minutes
  Vividity of Movement Imagery Questionnaire 2 will be used to assess the participant's imaging ability. Scores that can be obtained from the scale range between 16-80. High scores mean that the level of visual imagery is high; low scores mean that the level of visual imagery or visualization is low.

SECONDARY OUTCOMES:
Life Quality | 5 - 10 minutes
  The Pediatric Quality of Life Questionnaire of the International Quality of Living Scale for Children will be used to assess the quality of life of children and adolescents. Scores that can be obtained from the scale range between 0-100. High scores mean better condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No